CLINICAL TRIAL: NCT04537533
Title: Intraoperative Tranexamic Acid Infusion in Low Dose Versus in High Dose for Reducing Blood Loss and Its Effect on Postoperative Thromboembolic Complications in Radical Cystectomy Operations
Brief Title: Tranexamic Acid Infusion in Low Dose Versus in High Dose for Reducing Blood Loss in Radical Cystectomy Operations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Mohamed Abbas, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BRC
Record Dates: First submitted 2020-08-30; First posted 2020-09-03 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- first group (Experimental): 1st group (A) will include 30 patients: each one will receive 15mg/kg of I.V tranexemic acid as a bolus over 10 minutes (loading dose) then 10mg/kg/hour of I.V tranexemic acid as infusion all through the operation.
  Interventions: Drug: Tranexamic acid; Other: Normal saline
- second group (Active Comparator): 2nd group (B) will include 30 patients: : each one will receive 5mg/kg of I.V tranexemic acid as a bolus over 10 minutes (loading dose) then 1mg/kg/hour of I.V tranexemic acid as infusion all through the operation.
  Interventions: Drug: Tranexamic acid; Other: Normal saline
- Third group (Placebo Comparator): 3rd group (C){controlled group} will include 30 patients: each one will receive saline (placebo) injection and infusion all through the operation.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Tranexamic acid — Intraoperative infusion
  Arms: first group; second group
Other: Normal saline — intravenous infusion

SUMMARY:
Bladder cancer is one of the most common cancers of the genitourinary tract in adults, and its incidence distinctly increases with age . In almost two-thirds of cases, the disease is superficial at presentation and involves the mucosal and sub mucosal layers or the lamina propria of the bladder, whereas ∼20% to 30% of patients have muscle-invasive tumors. Superficial bladder cancer is treated by transurethral endoscopic resection, which can be followed by endovesical therapy for patients at risk of disease recurrence and progression . In contrast, muscle-invasive bladder cancer is generally treated by radical cystectomy with pelvic lymph node dissection and then creation of urinary diversion to create an alternate route for urine passage, which demonstrates 10-year recurrence-free survival rates of 50% to 59% and overall survival rates of ∼45% .

These major surgeries have a prolonged operative times and are associated with significant risk of complications including high risk of perioperative bleeding and subsequent need for blood transfusion with significant postoperative complications, which are reportedly in the range of 24% to 64% .

DETAILED DESCRIPTION:
Among individual surgeons at institutions that perform many procedures, median intraoperative blood loss is between 600 and 1700 mL. The incidence of at least one intraoperative blood transfusion is 9 to 67%, and the postoperative transfusion risk is at least 15%. Among cystectomy patients who receive transfusion, a median of 2 units of blood cells are given. Therefore, it is very important to establish surgical and anesthetic protocols aimed at minimizing intraoperative blood loss and subsequent blood transfusion requirements in order to improve postoperative outcomes.

Venous thromboembolism (VTE) in radical cystectomy can account for up to 22% of total deaths after surgery . In the bladder cancer literature, symptomatic thromboembolic events occur in up to 8.3% of patients , but subclinical deep vein thrombosis (DVT) rates can be as high as 24.4% when examining an ultrasonography (US)-screened population . In fact, undergoing a RC is a significant, independent risk factor on multivariable analysis for developing a deep venous thrombosis.

Lysine analog drugs are synthetic derivatives of the amino acid lysine that reversibly block lysine-binding sites on plasminogen molecules. This action prevents the conversion of plasminogen to plasmin, the active enzyme that degrades fibrin clots. Therefore, lysine analogs decrease the breakdown of clots and are considered anti-fibrinolytics. There are two commonly studied lysine analogs, tranexamic acid and epsilon-aminocaproic acid. Both of these drugs have been shown to decrease blood loss and blood transfusion need during some surgeries without a significant increase in adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 70 years old
* Gender: Males and females
* ASA grade I - II
* Patients undergoing radical cystectomy for bladder cancer regardless of tumor stage and histology.
* Patients who have undergone previous surgery, radiation, or chemotherapy may be included.
* All forms of urinary diversion are allowed

Exclusion Criteria:

* Patient refusal.
* Patient with allergy to tranexamic acid.
* Patients have thromboembolic disease (active or diagnosed within 1 year), such as deep vein thrombosis (DVT), pulmonary embolism (PE), cerebral thrombosis or MI.
* Pregnancy.
* Patients with hematuria.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Effect of low dose and high dose tranexemic acid infusion on Intraoperative blood loss . | within the first 15 days
  Estimated Blood Loss and perioperative need for blood transfusion within the first 15 days .

SECONDARY OUTCOMES:
Postoperative thromboembolic events | within the first 15 days
  Post operative complications as deep venous thrombosis, pulmonary embolism, MI, cerebral stroke, blurred vision and seizures within the first 15 days .

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Rhijn BW, Burger M, Lotan Y, Solsona E, Stief CG, Sylvester RJ, Witjes JA, Zlotta AR. Recurrence and progression of disease in non-muscle-invasive bladder cancer: from epidemiology to treatment strategy. Eur Urol. 2009 Sep;56(3):430-42. doi: 10.1016/j.eururo.2009.06.028. Epub 2009 Jun 26. PMID 19576682
- [Background] Parkin DM. The global burden of urinary bladder cancer. Scand J Urol Nephrol Suppl. 2008 Sep;(218):12-20. doi: 10.1080/03008880802285032. PMID 19054893
- [Background] Thompson E. Urological oncology in Europe. Research highlights from the XVIIth congress of the European Association of Urology, Birmingham, UK, February 23-26, 2002. Drugs Today (Barc). 2002 Apr;38(4):221-34. No abstract available. PMID 12532191
- [Background] Meyer JP, Blick C, Arumainayagam N, Hurley K, Gillatt D, Persad R, Fawcett D. A three-centre experience of orthotopic neobladder reconstruction after radical cystectomy: revisiting the initial experience, and results in 104 patients. BJU Int. 2009 Mar;103(5):680-3. doi: 10.1111/j.1464-410X.2008.08204.x. Epub 2008 Dec 2. PMID 19076133
- [Background] Cookson MS, Chang SS, Wells N, Parekh DJ, Smith JA Jr. Complications of radical cystectomy for nonmuscle invasive disease: comparison with muscle invasive disease. J Urol. 2003 Jan;169(1):101-4. doi: 10.1016/S0022-5347(05)64045-1. PMID 12478113
- [Background] Lawrentschuk N, Colombo R, Hakenberg OW, Lerner SP, Mansson W, Sagalowsky A, Wirth MP. Prevention and management of complications following radical cystectomy for bladder cancer. Eur Urol. 2010 Jun;57(6):983-1001. doi: 10.1016/j.eururo.2010.02.024. Epub 2010 Feb 26. PMID 20227172
- [Background] Lowrance WT, Rumohr JA, Chang SS, Clark PE, Smith JA Jr, Cookson MS. Contemporary open radical cystectomy: analysis of perioperative outcomes. J Urol. 2008 Apr;179(4):1313-8; discussion 1318. doi: 10.1016/j.juro.2007.11.084. Epub 2008 Mar 4. PMID 18289578
- [Background] Chang SS, Smith JA Jr, Wells N, Peterson M, Kovach B, Cookson MS. Estimated blood loss and transfusion requirements of radical cystectomy. J Urol. 2001 Dec;166(6):2151-4. PMID 11696725
- [Background] Shabsigh A, Korets R, Vora KC, Brooks CM, Cronin AM, Savage C, Raj G, Bochner BH, Dalbagni G, Herr HW, Donat SM. Defining early morbidity of radical cystectomy for patients with bladder cancer using a standardized reporting methodology. Eur Urol. 2009 Jan;55(1):164-74. doi: 10.1016/j.eururo.2008.07.031. Epub 2008 Jul 18. PMID 18675501
- [Background] Novara G, De Marco V, Aragona M, Boscolo-Berto R, Cavalleri S, Artibani W, Ficarra V. Complications and mortality after radical cystectomy for bladder transitional cell cancer. J Urol. 2009 Sep;182(3):914-21. doi: 10.1016/j.juro.2009.05.032. Epub 2009 Jul 17. PMID 19616246
- [Background] Hautmann RE, de Petriconi RC, Volkmer BG. Lessons learned from 1,000 neobladders: the 90-day complication rate. J Urol. 2010 Sep;184(3):990-4; quiz 1235. doi: 10.1016/j.juro.2010.05.037. PMID 20643429
- [Background] Quek ML, Stein JP, Daneshmand S, Miranda G, Thangathurai D, Roffey P, Skinner EC, Lieskovsky G, Skinner DG. A critical analysis of perioperative mortality from radical cystectomy. J Urol. 2006 Mar;175(3 Pt 1):886-9; discussion 889-90. doi: 10.1016/S0022-5347(05)00421-0. PMID 16469572
- [Background] Clement C, Rossi P, Aissi K, Barthelemy P, Guibert N, Auquier P, Ragni E, Rossi D, Frances Y, Bastide C. Incidence, risk profile and morphological pattern of lower extremity venous thromboembolism after urological cancer surgery. J Urol. 2011 Dec;186(6):2293-7. doi: 10.1016/j.juro.2011.07.074. Epub 2011 Oct 20. PMID 22014814
- [Background] Nilsson IM. Clinical pharmacology of aminocaproic and tranexamic acids. J Clin Pathol Suppl (R Coll Pathol). 1980;14:41-7. No abstract available. PMID 7000846